CLINICAL TRIAL: NCT00902057
Title: Effect of Desmopressin on Platelet Dysfunction Associated With Mild Hypothermia in Healthy Volunteers
Brief Title: Desmopressin for Bleeding Related to Low Body Temperature
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Dr Kwok Fu Jacobus Ng, Department of Anaesthesiology, the Univeristy of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW 09-088
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Hypothermia Induced Impairment of Primary Haemostasis
MeSH Terms: interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- desmopressin 1.5 (Active Comparator)
  Interventions: Drug: desmopressin
- desmopressin 3 (Active Comparator)
  Interventions: Drug: desmopressin
- desmopressin 15 (Active Comparator)
  Interventions: Drug: desmopressin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: desmopressin — single desmopressin subcutaneous injection, 1.5mcg
  Arms: desmopressin 1.5
Drug: desmopressin — single desmopressin subcutaneous injection, 3mcg
  Arms: desmopressin 3
Drug: desmopressin — single desmopressin subcutaneous injection, 15mcg
  Arms: desmopressin 15
Drug: placebo — saline subcutaneous
  Arms: placebo

SUMMARY:
To study, with a prospective randomised controlled design, whether the subcutaneous administration of the haemostatic drug desmopressin, may improve the impairment of primary haemostasis due to mildly decreased temperature.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers

Exclusion Criteria:

1. Any known platelet or coagulation disorder.
2. Pregnant or lactating women.
3. Known chronic liver or renal disease.
4. Coronary artery, carotid artery or peripheral artery disease
5. Recent history of taking antiplatelet drugs, anticoagulants or herbal preparations.
6. Smoker or alcohol user
7. Mentally incapable of providing informed consent
8. Students or junior staff members who had direct working relationship with the PI

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
closure time on PFA-100 | 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong, China